CLINICAL TRIAL: NCT01064284
Title: Inhibitor Development in Previously Untreated Patients (PUPs) or Minimally Blood Component-Treated Patients (MBCTPs) When Exposed to Plasma-derived Von Willebrand Factor-Containing Factor VIII (VWF/FVIII) Concentrates and to Recombinant Factor VIII (rFVIII) Concentrates: An Independent, International, Multicentre, Prospective, Controlled, Randomised, Open Label, Clinical Trial
Brief Title: Survey of Inhibitors in Plasma-Product Exposed Toddlers
Acronym: SIPPET
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fondazione Angelo Bianchi Bonomi (Other)
Collaborators: Sintesi Research Srl (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ABB - 09 - 001; 2009-011186-88 (EudraCT Number)
Record Dates: First submitted 2010-02-04; First posted 2010-02-08 (Estimated); Results first posted 2017-04-07 (Actual); Last update posted 2017-08-25 (Actual); Status verified 2017-07

CONDITIONS: Hemophilia A
Keywords: Hemophilia A; Factor VIII inhibitors; vWF/FVIII; rFVIII
MeSH Terms: conditions — Hemophilia A | interventions — factor VIII, von Willebrand factor drug combination; recombinant FVIII, sugar formulated; Factor VIII

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PLASMA DERIVED Factor VIII (Active Comparator): Plasma-derived vWF/FVIII
  Interventions: Drug: PLASMA DERIVED Factor VIII
- rFVIII (Active Comparator): Recombinant FVIII
  Interventions: Drug: Recombinant FVIII

INTERVENTIONS:
Drug: PLASMA DERIVED Factor VIII — Maximum dosage : 50IU per kilo. 2-3 times per week or on demand during acute episode of bleeding
  Other Names: ALPHANATE
  Arms: PLASMA DERIVED Factor VIII
Drug: Recombinant FVIII — Maximum dosage : 50IU per kilo. 2-3 times per week or on demand during acute episode of bleeding
  Other Names: ADVATE
  Arms: rFVIII

SUMMARY:
The primary objective of the study is to assess the immunogenicity of VWF/FVIII and of rFVIII concentrates by determining the frequency of inhibitor development in previously untreated patients (PUPs) or minimally blood component-treated (MBCTPs) in the first 50 EDs or in the first 3 years from enrollment, whichever occurs first.

.

DETAILED DESCRIPTION:
Patients meeting the enrollment criteria will be consecutively enrolled at each participating centre, randomized to be treated exclusively with a single FVIII product either plasma-derived or recombinant, and followed up until inhibitor development or until 50 exposure days (EDs) or 3 years from enrolment have elapsed, whichever comes first. Study products, belonging to the class of rFVIII concentrates and to the class of plasma-derived VWF/FVIII concentrates, will be provided for free to the patients for all the duration of the study

ELIGIBILITY:
Inclusion Criteria:

* Male subjects
* Any ethnicity
* Age <6 years
* Severe haemophilia A (FVIII:C <1%), as confirmed at enrolment by the central laboratory.

  o Those patients diagnosed locally as severe but subsequently found to have FVIII levels >= 1% on testing at the central laboratory will be separately recorded in the screening list.
* Previously untreated (0 EDs to any FVIII concentrates or blood products) or minimally treated (<5 EDs) with blood components, namely whole blood, fresh frozen plasma, packed red blood cells, platelets or cryoprecipitate.

  o Patients not meeting these criteria will be separately recorded in the screening list.
* Negative inhibitor measurement at both local and central laboratory at screening
* Ability to comply with study requirements
* Signed informed consent of legal tutors o Patients who will not accept to enter into the study or to be randomized will be separately recorded.

Exclusion Criteria:

* Previous history of FVIII inhibitor
* Other congenital or acquired bleeding defects
* Plasma FVIII level >= 1%, as assayed at the central laboratory

  o Those patients originally diagnosed locally as severe but subsequently found to have FVIII levels ranging from 1% to 2% on testing at the central laboratory will be separately recorded in the screening list.
* Concomitant congenital or acquired immunodeficiency
* Concomitant treatment with systemic immunosuppressive drugs
* Concomitant treatment with any investigational drug

Ages: 1 Minute to 6 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 303 (Actual)
Dates: Start 2010-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pier M. Mannucci, Professor, Principal Investigator — Fondazione Ca' Granda Ospedale Maggiore Policlinico Milano; Flora Peyvandi, Professor, Principal Investigator — Fondazione Ca' Granda Ospedale Maggiore Policlinico Milano
Locations (48):
- United States (10):
  - City of Hope National Medical Center, Duarte, California
  - Children's Hospital Los Angeles (CHLA), Los Angeles, California
  - Hemophilia and Thrombosis CenterUniversity of Colorado Denver - Anschutz Aurora, Aurora, Colorado
  - Rush Hemophilia & Trombophilia Center - Rush University Medical Center, Chicago, Illinois
  - Louisiana Center for Bleeding and Clotting Disorders, Tulane University Medical Center, New Orleans, Louisiana
  - University of Mississippi Medical Center, Division of pediatric Hematology/Oncology, Jackson, Mississippi
  - Children's Mercy Hospital, Kansas City, Missouri
  - Hemophilia Treatment Center of Las Vegas, Las Vegas, Nevada
  - MeritCare Roger Maris Cancer Center, Pediatric Oncology, Fargo, North Dakota
  - Cook Children's Medical Center, Fort Worth, Texas
- Argentina (2):
  - Hospital de Ninos Sor Maria Ludovica La Plata Servicio de Hematologia, La Plata, Buenos Aires
  - Fundacion de la Hemofilia, Buenos Aires
- Austria (2):
  - Landes- Frauen- und Kinderklinik Linz Abteilung für Kinder- und Jugendheilkunde, Linz
  - Medizinische Universität Wien, Dept. Paediatrics, Vienna
- Brazil (2):
  - Centro de Pesquisa Clinica HEMORIO - Instituto Estadual de Hematologia Arthur de Siqueira Cavalcanti, Rio de Janeiro
  - Centro de Hematologia e Hemoterapia do e.s - Hemoes, Vitória
- Chile (2):
  - Hospital de Niños Dr. Luis Calvo Mackenna Centro Hemofílico, Santiago
  - Centro de Hemofilicos del Hospital de Niños Roberto del Rio Instituto de Investigaciones Hematologicas, Santiago
- Egypt (2):
  - Paediatric Haematology department, Cairo University Pediatric Hospital, Cairo
  - Faculty of Medicine Ain Shams University Department Pediatrics, Cairo
- India (10):
  - Centre for Blood Disorders, Chennai
  - St. John's Medical College & Hospital, Karnataka
  - Kasturba Medical College, Manipal University, Karnataka
  - Karnataka Hemophilia Care and Hematology Research Center, Karnataka
  - Kerala Institute of Medical Science (KIMS), Kerala
  - Lokmanya TilakMunicipal Medical College &General Hospital - Sion, Mumbai
  - All India Institute of Medical Sciences Department of Haematology, New Delhi
  - Sir Ganga Ram Hospital, New Delhi
  - Sahyadri Speciality Hospital, Pune
  - Jehangir Clinical Development Centre, Department of Haematology, Jehangir Hospital Premises, Pune
- Iran (2):
  - Hemophilia Center - Hematoogy & Oncology Dept. Shiraz University of Medical Science Ayatollah Dastgheib Hospital, Shiraz
  - Comprehensive Care Center for Children with Hemophilia Mofid Children Hospital, Tehran
- Italy (3):
  - Centro Emofilia e Trombosi "Angelo Bianchi Bonomi" Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico di Milano - Italy, Milan
  - Clinica Medica II - Azienda Ospedaliera di Padova - Centro Emofilia di Padova, Padua
  - Ematologia- UO Diagnostica Speciale e Terapia delle Malattie dell'Emostasi e della Trombosi- Università Sapienza - Policlinico Umberto I, Rome
- Mexico (5):
  - Unidad Medica de Alta Especialidad (UMAE), Hospital de Pediatria. Centro Medico Nacional de Occidente Istituto Mexicano del Seguro Social, Jalisco
  - Instituto Nacional de Pediatria, México D.F.
  - Hospital Infantil de Mexico Federico Gomez, México, D.F.
  - Hospital Universitario Dr. Josè Eleuterio Gonzalez de la UANL, NL. Mexico, Monterrey
  - Hospital de Especialidades UMAE Istituto Mexicano del Seguro Social (IMSS), Monterrey (Nuevo Leòn)
- Kinf Faisal Specilist Hospital and Research Center, Riyadh, Saudi Arabia
- Haemophilia Comprehensive Care Clinic, Area 454, Charlotte Maxeke Johannesburg Academic Hospital, Parktown, South Africa
- Spain (3):
  - Hospital Regional Universitario Carlos Haya, Málaga
  - Hospital Universitario Virgen del Rocio Unidad de Hemofilia, Seville
  - Hospital Universitario La Fe Unidad Coagulopatias Congenitas, Valencia
- Turkey (Türkiye) (3):
  - Cukurova Universitesi, Tip Fakultesi Pediatrik Hematoloji B.D., Adana
  - Ege Üniversitesi Tip Fakültesi Cocuk Sağliği ve Hastalikari Anabilim Dali Pediatrik Hematoloji Bilim Dali, Bornova/Izmir
  - Istanbul Üniversitesi Cerrahpaşa Tip Fakültesi Pediatrik Hematoloji B.D., Istanbul

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) are available to other researchers through the publication of an article.

REFERENCES:
- [Background] Addiego J, Kasper C, Abildgaard C, Hilgartner M, Lusher J, Glader B, Aledort L. Frequency of inhibitor development in haemophiliacs treated with low-purity factor VIII. Lancet. 1993 Aug 21;342(8869):462-4. doi: 10.1016/0140-6736(93)91593-b. PMID 8102429
- [Background] Amano K, Arai M, Koshihara K, Suzuki T, Kagawa K, Nishida Y, Fukutake K. Autoantibody to factor VIII that has less reactivity to factor VIII/von Willebrand factor complex. Am J Hematol. 1995 Aug;49(4):310-7. doi: 10.1002/ajh.2830490409. PMID 7639276
- [Background] Auerswald G, Spranger T, Brackmann HH. The role of plasma-derived factor VIII/von Willebrand factor concentrates in the treatment of hemophilia A patients. Haematologica. 2003 Jun;88(6):EREP05. PMID 12826531
- [Background] Chalmers EA, Brown SA, Keeling D, Liesner R, Richards M, Stirling D, Thomas A, Vidler V, Williams MD, Young D; Paediatric Working Party of UKHCDO. Early factor VIII exposure and subsequent inhibitor development in children with severe haemophilia A. Haemophilia. 2007 Mar;13(2):149-55. doi: 10.1111/j.1365-2516.2006.01418.x. PMID 17286767
- [Background] Courter SG, Bedrosian CL. Clinical evaluation of B-domain deleted recombinant factor VIII in previously untreated patients. Semin Hematol. 2001 Apr;38(2 Suppl 4):52-9. doi: 10.1016/s0037-1963(01)90109-x. PMID 11449336
- [Background] Dasgupta S, Repesse Y, Bayry J, Navarrete AM, Wootla B, Delignat S, Irinopoulou T, Kamate C, Saint-Remy JM, Jacquemin M, Lenting PJ, Borel-Derlon A, Kaveri SV, Lacroix-Desmazes S. VWF protects FVIII from endocytosis by dendritic cells and subsequent presentation to immune effectors. Blood. 2007 Jan 15;109(2):610-2. doi: 10.1182/blood-2006-05-022756. Epub 2006 Sep 19. PMID 16985172
- [Background] Ehrenforth S, Kreuz W, Scharrer I, Linde R, Funk M, Gungor T, Krackhardt B, Kornhuber B. Incidence of development of factor VIII and factor IX inhibitors in haemophiliacs. Lancet. 1992 Mar 7;339(8793):594-8. doi: 10.1016/0140-6736(92)90874-3. PMID 1347102
- [Background] Goudemand J, Rothschild C, Demiguel V, Vinciguerrat C, Lambert T, Chambost H, Borel-Derlon A, Claeyssens S, Laurian Y, Calvez T; FVIII-LFB and Recombinant FVIII study groups. Influence of the type of factor VIII concentrate on the incidence of factor VIII inhibitors in previously untreated patients with severe hemophilia A. Blood. 2006 Jan 1;107(1):46-51. doi: 10.1182/blood-2005-04-1371. Epub 2005 Sep 15. PMID 16166584
- [Background] Gouw SC, van der Bom JG, Auerswald G, Ettinghausen CE, Tedgard U, van den Berg HM. Recombinant versus plasma-derived factor VIII products and the development of inhibitors in previously untreated patients with severe hemophilia A: the CANAL cohort study. Blood. 2007 Jun 1;109(11):4693-7. doi: 10.1182/blood-2006-11-056317. Epub 2007 Jan 11. PMID 17218379
- [Background] Gringeri A, Mantovani LG, Scalone L, Mannucci PM; COCIS Study Group. Cost of care and quality of life for patients with hemophilia complicated by inhibitors: the COCIS Study Group. Blood. 2003 Oct 1;102(7):2358-63. doi: 10.1182/blood-2003-03-0941. Epub 2003 Jun 19. PMID 12816859
- [Background] Gringeri A, Monzini M, Tagariello G, Scaraggi FA, Mannucci PM; Emoclot15 Study Members. Occurrence of inhibitors in previously untreated or minimally treated patients with haemophilia A after exposure to a plasma-derived solvent-detergent factor VIII concentrate. Haemophilia. 2006 Mar;12(2):128-32. doi: 10.1111/j.1365-2516.2006.01201.x. PMID 16476086
- [Background] Guerois C, Laurian Y, Rothschild C, Parquet-Gernez A, Duclos AM, Negrier C, Vicariot M, Fimbel B, Fressinaud E, Fiks-Sigaud M, et al. Incidence of factor VIII inhibitor development in severe hemophilia A patients treated only with one brand of highly purified plasma-derived concentrate. Thromb Haemost. 1995 Feb;73(2):215-8. PMID 7792732
- [Background] Kreuz W, Gill JC, Rothschild C, Manco-Johnson MJ, Lusher JM, Kellermann E, Gorina E, Larson PJ; International Kogenate-FS Study Group. Full-length sucrose-formulated recombinant factor VIII for treatment of previously untreated or minimally treated young children with severe haemophilia A: results of an international clinical investigation. Thromb Haemost. 2005 Mar;93(3):457-67. doi: 10.1160/TH03-10-0643. PMID 15735795
- [Background] Lorenzo JI, Lopez A, Altisent C, Aznar JA. Incidence of factor VIII inhibitors in severe haemophilia: the importance of patient age. Br J Haematol. 2001 Jun;113(3):600-3. doi: 10.1046/j.1365-2141.2001.02828.x. PMID 11380444
- [Background] Lusher JM, Arkin S, Abildgaard CF, Schwartz RS. Recombinant factor VIII for the treatment of previously untreated patients with hemophilia A. Safety, efficacy, and development of inhibitors. Kogenate Previously Untreated Patient Study Group. N Engl J Med. 1993 Feb 18;328(7):453-9. doi: 10.1056/NEJM199302183280701. PMID 8421474
- [Background] O'Brien PC, Fleming TR. A multiple testing procedure for clinical trials. Biometrics. 1979 Sep;35(3):549-56. PMID 497341
- [Background] Qadura M, Waters B, Burnett E, Chegeni R, Othman M, Lillicrap D. Investigating the mechanisms underlying FVIII antibody production in hemophilic mice following recombinant and plasma-derived FVIII infusion. Blood (ASH Annual Meeting Abstracts) 2008; 112: abstract #237.
- [Background] Rothschild C, Laurian Y, Satre EP, Borel Derlon A, Chambost H, Moreau P, Goudemand J, Parquet A, Peynet J, Vicariot M, Beurrier P, Claeyssens S, Durin A, Faradji A, Fressinaud E, Gaillard S, Guerin V, Guerois C, Pernod G, Pouzol P, Schved JF, Gazengel C. French previously untreated patients with severe hemophilia A after exposure to recombinant factor VIII : incidence of inhibitor and evaluation of immune tolerance. Thromb Haemost. 1998 Nov;80(5):779-83. PMID 9843171
- [Background] Scharrer I, Ehrlich HJ. Reported inhibitor incidence in FVIII PUP studies: comparing apples with oranges? Haemophilia. 2004 Mar;10(2):197-8. doi: 10.1111/j.1365-2516.2004.00887.x. No abstract available. PMID 14962213
- [Background] Schimpf K, Schwarz P, Kunschak M. Zero incidence of inhibitors in previously untreated patients who received intermediate purity factor VIII concentrate or factor IX complex. Thromb Haemost. 1995 Mar;73(3):553-5. No abstract available. PMID 7667845
- [Background] Strauss T, Lubetsky A, Ravid B, Bashari D, Luboshitz J, Lalezari S, Misgav M, Martinowitz U, Kenet G. Recombinant factor concentrates may increase inhibitor development: a single centre cohort study. Haemophilia. 2011 Jul;17(4):625-9. doi: 10.1111/j.1365-2516.2010.02464.x. Epub 2011 Feb 7. PMID 21299743
- [Background] Waters B, Qadura M, Burnett E, Chegeni R, Labelle A, Thompson P, Hough C, Lillicrap D. Anti-CD3 prevents factor VIII inhibitor development in hemophilia A mice by a regulatory CD4+CD25+-dependent mechanism and by shifting cytokine production to favor a Th1 response. Blood. 2009 Jan 1;113(1):193-203. doi: 10.1182/blood-2008-04-151597. Epub 2008 Sep 24. PMID 18815284
- [Background] Wight J, Paisley S. The epidemiology of inhibitors in haemophilia A: a systematic review. Haemophilia. 2003 Jul;9(4):418-35. doi: 10.1046/j.1365-2516.2003.00780.x. PMID 12828678
- [Derived] Rosendaal FR, Palla R, Garagiola I, Mannucci PM, Peyvandi F; SIPPET Study Group. Genetic risk stratification to reduce inhibitor development in the early treatment of hemophilia A: a SIPPET analysis. Blood. 2017 Oct 12;130(15):1757-1759. doi: 10.1182/blood-2017-06-791756. Epub 2017 Aug 2. PMID 28768627
- [Derived] Peyvandi F, Mannucci PM, Garagiola I, El-Beshlawy A, Elalfy M, Ramanan V, Eshghi P, Hanagavadi S, Varadarajan R, Karimi M, Manglani MV, Ross C, Young G, Seth T, Apte S, Nayak DM, Santagostino E, Mancuso ME, Sandoval Gonzalez AC, Mahlangu JN, Bonanad Boix S, Cerqueira M, Ewing NP, Male C, Owaidah T, Soto Arellano V, Kobrinsky NL, Majumdar S, Perez Garrido R, Sachdeva A, Simpson M, Thomas M, Zanon E, Antmen B, Kavakli K, Manco-Johnson MJ, Martinez M, Marzouka E, Mazzucconi MG, Neme D, Palomo Bravo A, Paredes Aguilera R, Prezotti A, Schmitt K, Wicklund BM, Zulfikar B, Rosendaal FR. A Randomized Trial of Factor VIII and Neutralizing Antibodies in Hemophilia A. N Engl J Med. 2016 May 26;374(21):2054-64. doi: 10.1056/NEJMoa1516437. PMID 27223147
- See also: The official web site of the SIPPET Study — http://sippetstudy.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 303 boys were assessed for eligibility, 39 were excluded, therefore, of those 303, only 264 patients underwent randomization. Of these 264, only 251 were analyzed.
Groups:
- pd vWF/FVIII: Plasma-derived vWF/FVIII
  PLASMA DERIVED Factor VIII: Maximum dosage : 50IU per kilo. 2-3 times per week or on demand during acute episode of bleeding
Period: Overall Study
Arm/Group | pd vWF/FVIII | rFVIII
Started | 125 (Taking into account the analyzed patients only) | 126 (Taking into account the analyzed patients only)
Completed | 107 | 109
Not Completed | 18 | 17

BASELINE CHARACTERISTICS:
Population: It is considered as "Baseline Analysis Population" only the one actually analyzed at the end of the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | pd vWF/FVIII | rFVIII | Total
Number analyzed (Participants) | 125 | 126 | 251
Age, Continuous [Mean (Standard Deviation); unit: months] — Age at first treatment
  months | 19.1 (14.3) | 21.3 (16.3) | 20.2 (21.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 125 | 126 | 251
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 41 | 43 | 84
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 2 | 7
  White | 39 | 45 | 84
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 40 | 36 | 76
Region of Enrollment [Number; unit: participants]
  Argentina | 2 | 0 | 2
  Austria | 2 | 2 | 4
  Brazil | 2 | 2 | 4
  Chile | 1 | 3 | 4
  Egypt | 38 | 37 | 75
  India | 40 | 43 | 83
  Iran | 14 | 18 | 32
  Italy | 5 | 4 | 9
  Mexico | 4 | 2 | 6
  Saudi Arabia | 1 | 0 | 1
  South Africa | 2 | 2 | 4
  Spain | 3 | 3 | 6
  Turkey | 2 | 1 | 3
  United States | 9 | 9 | 18
Mutation Status [Number; unit: participants] — Population: There were no cells or DNA available for 17 patients.
  participants
    Non-null mutation: number analyzed (Participants) | 117 | 117 | 234
    Non-null mutation | 16 | 21 | 37
    Null mutation: number analyzed (Participants) | 117 | 117 | 234
    Null mutation | 101 | 96 | 197
Treatment Regimen [Number; unit: participants]
  On-demand | 61 | 56 | 117
  Standard prophylaxis | 21 | 19 | 40
  Modified prophylaxis | 43 | 51 | 94

OUTCOME MEASURES:

1. Primary Outcome: To Assess the Immunogenicity of Plasma Derived VWF/FVIII and rFVIII Concentrates by Determining the Frequency of Inhibitor Development in the First 50 EDs or in the First 3 Years From Enrolment, Whichever Comes First in PUPs and MBCTs
Description: Expressed with the numebr of patients for each group who developed FVIII inhibitors.
  PUPs: Previously Untreated Patients MBCTPs: Minimally Blood Component-Treated Patients
Time Frame: During the first 50 exposure days or first 3 years of enrollment, whichever occurs first
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | pd vWF/FVIII | rFVIII
Number analyzed (Participants) | 125 | 126
participants | 29 [18.4 to 35.2] | 47 [34.7 to 54.3]

2. Secondary Outcome: To Evaluate the Anamnestic Response of Inhibitor Patients
Time Frame: During the first 50 exposure days or first 3 years of enrollment, whichever occurs first
Population: Data were not collected and the Outcome will never be analyzed.
Arm/Group | PLASMA DERIVED Factor VIII | rFVIII
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: To Evaluate the Frequency of Transient Inhibitors
Description: Number of participants for each group who developed transient inhibitors (this means, those inhibitors which disappeared spontaneously within 6 months without immunotolerance treatment).
Time Frame: In the 6 months after inhibitor development
Population: Data at 6-month follow-up were missing for two patients assigned to plasma- derived factor VIII and three patients assigned to recombinant factor VIII.
Measure: Number; unit: participants
Arm/Group | pd vWF/FVIII | rFVIII
Number analyzed (Participants) | 123 | 123
participants | 7 | 12

4. Secondary Outcome: To Evaluate the Modality of Occurrence of Inhibitors (Number of EDs)
Description: Number of EDs: Number of Exposure Days (EDs) after which the inhibitors develop
Time Frame: During the first 50 exposure days or first 3 years of enrollment, whichever occurs first
Measure: Median (Full Range); unit: Exposure days
Arm/Group | pd vWF/FVIII | rFVIII
Number analyzed (Participants) | 125 | 126
Exposure days | 8 [3 to 33] | 8 [2 to 38]

5. Secondary Outcome: To Evaluate the Modality of Occurrence of Inhibitors (Titre at Onset)
Description: Inhibitor Titre at Onset
Time Frame: During 6 months of observation, from the inhibitor occurrence
Measure: Median (Full Range); unit: Bethesda Units
Arm/Group | pd vWF/FVIII | rFVIII
Number analyzed (Participants) | 125 | 126
Bethesda Units | 12 [0.8 to 1100] | 16.3 [0.7 to 1850]

6. Secondary Outcome: To Evaluate Clinical Factors Potentially Associated to Inhibitor Development
Time Frame: During the first 50 exposure days or first 3 years of enrollment, whichever occurs first
Population: Data were not collected and the Outcome will never be analyzed
Arm/Group | pd vWF/FVIII | rFVIII
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: To Evaluate Laboratory Factors Potentially Associated to Inhibitor Development
Time Frame: During the first 50 exposure days or first 3 years of enrollment, whichever occurs first
Population: Data were not collected and the Outcome will never be analyzed
Arm/Group | pd vWF/FVIII | rFVIII
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: To Evaluate the Incidence of All Other Adverse Events Related and Not Related to the Products Used
Time Frame: During the first 50 exposure days or first 3 years of enrollment, whichever occurs first
Population: Data were not collected and the Outcome will never be analyzed
Arm/Group | pd vWF/FVIII | rFVIII
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 5 years
Description: Systematic Assessment has been applied through the use of a specific routinary questions focusing on averse events and a patient's diary.
Arm/Group | pd vWF/FVIII | rFVIII
Serious Adverse Events (participants affected / at risk) | 20/133 | 13/131
Other Adverse Events (participants affected / at risk) | 95/133 | 86/131
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | pd vWF/FVIII (N=133) | rFVIII (N=131)
Abdominal wall haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) — Leading to death
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Circumcision (Surgical and medical procedures) | 1 (1) | 0 (0)
Epidural Haemorrage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 3 (3) — In one case (pd vWF/FVIII) leading to death
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Head Injury (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0)
Hemiplegia (Nervous system disorders) | 1 (1) | 0 (0)
Hepatomegaly (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hypersomnia (Nervous system disorders) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lower Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Poor venous access (Vascular disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Speech disorder developmental (Nervous system disorders) | 1 (1) | 0 (0)
Status epilepticus (Nervous system disorders) | 0 (0) | 1 (1)
Subcutaneous haematoma (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Talipes correction (Surgical and medical procedures) | 0 (0) | 1 (1)
Torticollis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Vessel puncture site haemorrhage (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | pd vWF/FVIII (N=133) | rFVIII (N=131)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 8 (8)
Bronchitis (Infections and infestations) | 7 (8) | 5 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (12) | 9 (34)
Diarrhoea (Gastrointestinal disorders) | 6 (8) | 7 (9)
Nasopharyngitis (Infections and infestations) | 16 (19) | 10 (42)
Pharyngitis (Infections and infestations) | 3 (9) | 8 (10)
Pyrexia (General disorders) | 22 (37) | 16 (37)
Upper respiratory tract infection (Infections and infestations) | 11 (17) | 9 (12)
Viral infection (Infections and infestations) | 8 (13) | 6 (9)
Vomiting (Gastrointestinal disorders) | 8 (11) | 8 (9)

LIMITATIONS AND CAVEATS:
Enrollment early termination,because on September2014 WFH stated:with other safe clotting-factor concentrates available,consider not to use Kogenate FS/Helixate NexGen(CSL Behring)for newly diagnosed Severe Haemophilia A patients not treated before.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No